CLINICAL TRIAL: NCT04423172
Title: Safety, Efficacy and Operability of Using the New Tissue Containment System With Hard Pipes Which Can Assemble With Detachable Trocars Seamlessly for Tissue Removal During Laprascopic Hysterectomy
Brief Title: Safety, Efficacy and Operability of Using the New Tissue Containment System During Laprascopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jing Liang (Other)
Responsible Party: Sponsor-Investigator, Jing Liang, professor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTCS-LH
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Gynecologic Surgery
Keywords: morcellation; laparoscopic surgery; hysterectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using the New Tissue Containment System group (Experimental): using the new tissue containment system during Laparoscopic Hysterectomy. The divice is a soft specimen bag in which the uterus tissue is sealed and quickly morcellation and removed through vagina. The divice is named the new tissue containment system.
  Interventions: Device: the new tissue containment system
- Open group (No Intervention): Without using any procteciton system during Laprascopic Hysterectomy.

INTERVENTIONS:
Device: the new tissue containment system — Using the new tissue containment system during Laparoscopic hysterectomy. The divice is a soft specimen bag in which the uterus tissue is sealed and quickly morcellation and removed through vagina. The divice is named the new tissue containment system.
  Arms: Using the New Tissue Containment System group

SUMMARY:
The study is designed to evaluate the safety, operability and efficacy of performing the new tissue containment system during laparoscopic hysterectomy. Pre- and perimenopausal women undergoing laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and Peri-menopausal woman patient age 18-65 years
* Women with fibroids, adenomyosis, and endometrial hyperplasia and indication for laparoscopic hysterectomy.
* Normal Pap smear result within one year
* The uterus is larger than 12 weeks of gestation
* The body mass index of the patients is 18.5-27.9kg/m2
* Signed informed consent form

Exclusion Criteria:

* Women with Known or suspected malignancy
* patients during pregnancy and lactation
* Known blood diseases, bleeding coagulation disease, any part of the active bleeding or bleeding tendency of the constitution of the patient
* Patients with known severe liver and kidney dysfunction;Liver function (ALT, AST) ≥ 2 times of normal upper limit, or renal function (Cr) ≥ normal upper limit
* Patients who are known to have participated in any other clinical trial within 3 months
* Patients who cannot sign informed consent
* Patients with acute stage infection of the reproductive system or other sites

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-16 (Estimated); Primary Completion 2021-06-16 (Estimated); Study Completion 2022-12-26 (Estimated)

PRIMARY OUTCOMES:
The exposure rate | approximately two years
  Exposure is defined as "disruption of the device (using dye leak testing or water testing) or visible tissue dissemination".

SECONDARY OUTCOMES:
Mean procedure time | Within one day after the surgery
  Mean procedure time will be measured by hour/minutes.
The probability of failure during in-bag morcellation procedure | approximately two years
  Failure is defined as the operator's inability to successfully insert and extract the device.
Estimated blood loss during operation | Within one day after the surgery
  Blood loss during operation will be measured by volume (mL)
Post-operative pain | Within one month after the surgery
  The patients' post-operative pain will be measured by The Visual Analog Score （VAS).The maximum value is 10 and the minimum is 0. The lower score means a better outcome.
Rate of intra- or post-operative complications | Three months after the surgery
  Intra or post complications rate (e.g. urinary, intestinal or nerve injury)
The Surgeon Task Load Index | Within one week after the surgery
  The Surgery Task Load Index will be measured by questionaire. The maximum value is 120 and the minimum is 0. The higher score means a worse outcome.
The Patients' life quality postoperative | One months after the surgery
  The patients' life quality will be measured by The World Health Organization's Quality of Life Questionnaire-Brief Version（WHOQOL-BREF).The maximum value is 120 and the minimum is 0. The higher score means a better outcome.

IPD SHARING:
Plan to Share IPD: Undecided
IPD will to be shared with other researchers after four years